CLINICAL TRIAL: NCT07182422
Title: Impact of Kremezin on Renal Recovery and Uremic Toxin Levels in Patients With Acute Kidney Disease
Brief Title: AST-120 (Kremezin®) for the Renal Protection and Attenuation of Decline in Acute Kidney Disease
Acronym: ASTRA-AKD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Conmed Pharmaceutical & Bio-Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202401872A3
Record Dates: First submitted 2025-09-04; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-05

CONDITIONS: Acute Kidney Disease; Acute Kidney Injury (AKI)
Keywords: Acute Kidney Disease (AKD); Acute Kidney Injury (AKI); Progression from AKI to CKD
MeSH Terms: conditions — Acute Kidney Injury | interventions — AST 120

STUDY DESIGN:
Intervention Model Description: 1. Experimental Group (AST-120 Treatment Group):
     * Drug: AST-120 (Kremezin®)
     * Dosage: 6 grams per day
     * Administration: Oral administration, in the form of 1 packet (2 grams) three times per day (TID)
     * Frequency: Three times daily, preferably with meals
     * Duration: 14 days of continuous treatment
     * Background Treatment: In addition to AST-120, participants will receive standard post-AKD care, including the avoidance of nephrotoxic agents and regular monitoring of renal function.
  2. Control Group (Standard Post-AKD Care Only):
     * Treatment: Participants will receive only standard post-AKD care, which involves:
     * Avoidance of nephrotoxic medications
     * Regular monitoring of renal function (e.g., serum creatinine and eGFR assessments)
     * Other supportive therapies as deemed necessary based on individual patient conditions
     * Duration: The control group will be monitored for the same 14-day period as the experimental group, with regular follow-ups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control (Standard Care Only) Intervention: Standard post-AKD care No AST-120
- Experimental (AST-120 + Standard Care) (Experimental): Intervention: AST-120 (Kremezin®) Dosage: 6 g/day (2 g TID, oral) Duration: 14 days Background treatment: Standard post-AKD care
  Interventions: Drug: AST-120 (Kremezin®)

INTERVENTIONS:
Drug: AST-120 (Kremezin®) — AST-120 (Kremezin®) Dosage: 6 g/day (2 g TID, oral) Duration: 14 days Background treatment: Standard post-AKD care
  Arms: Experimental (AST-120 + Standard Care)

SUMMARY:
The primary goal of this clinical trial is to evaluate the efficacy of AST-120 (Kremezin®) in combination with standard care in reducing the levels of protein-bound uremic toxins (PBUTs), specifically indoxyl sulfate (IS) and p-cresyl sulfate (p-CS), in patients with acute kidney disease (AKD). The trial aims to assess whether AST-120 can prevent further renal deterioration and slow the progression from AKD to chronic kidney disease (CKD) by mitigating the accumulation of PBUTs. Additionally, the study will investigate the potential of AST-120 to reduce the risk of CKD-associated complications, including cardiovascular disease, by reducing PBUT levels in AKD patients.

DETAILED DESCRIPTION:
Study Procedures：

1. Total Number of Subjects The total number of subjects planned for enrollment is 100.

The study will include two groups:

1. Experimental Group: 50 patients receiving AST-120 (6g/day) in combination with standard post-AKD care.
2. Control Group: 50 patients receiving only standard post-AKD care. The sample size is determined based on the statistical power needed to detect a significant difference in the primary endpoint (percentage changes in IS levels), with consideration for potential dropout rates. The evaluable number is estimated to be close to 90, allowing for a 10% dropout rate, making the enrolled number 100.

2. Interventions, Procedures, and Tests for Each Group

Subjects will undergo the following interventions, procedures, and tests according to the schedule:

1. Baseline (Day 0):

   - Demographic data collection.
   * Blood tests for serum creatinine, eGFR, IS, p-CS, and urinary albumin-to-creatinine ratio (UACR).
   * Randomization into experimental or control groups.
2. Treatment Period (Day 1-14):

   * Experimental Group: Receive AST-120 (6g/day, divided into three doses per day).
   * Control Group: Standard post-AKD care only.
   * Both groups will undergo regular clinical assessments and adverse event monitoring.
3. Day 14:

   * Blood tests for IS, p-CS, serum creatinine, eGFR, and UACR.
   * Follow-up (Day 90 and Day 180):
   * Assess eGFR, serum creatinine, UACR.
   * Monitor for major adverse kidney events (MAKE) and major adverse cardiovascular events (MACE).

     3. Trial Procedure Timeline

The trial procedure follows this timeline:

1. Day 0: Baseline measurements and randomization.
2. Day 1-14: Treatment phase (AST-120 administration or standard care).
3. Day 14: Blood tests and assessment of treatment efficacy.
4. Day 90 and Day 180: Follow-up visits for MAKE and MACE assessments, and blood tests for kidney function.

4. Specimen Collection and Processing

1. Specimen: Blood samples will be collected on Day 0 (baseline), Day 14 (end of treatment), Day 90, and Day 180 (follow-up).
2. Transport and Storage: Specimens will be transported to the laboratory within the hospital for immediate processing. They will be stored in a temperature-controlled facility if needed.
3. Processing: Blood samples will undergo centrifugation for serum separation. Serum will be used for measuring IS, p-CS, serum creatinine, and other biomarkers.
4. Analysis: The following tests will be performed:

   * IS and p-CS levels.
   * Serum creatinine and eGFR.
   * UACR.

     5. Clinical Data Collection and Questionnaires

Clinical data collected will include:

1. Demographic data (age, sex, medical history).
2. Lab results for IS, p-CS, creatinine, eGFR, UACR. No specific questionnaires will be used for this study.

ELIGIBILITY:
Inclusion/Exclusion Criteria： Inclusion criteria

1. Age between 18 and 80 years.
2. Diagnosis of acute kidney disease (AKD) during hospitalization, with AKD stage 2 or 3 according to the KDIGO-AKD criteria, defined by an increase in serum creatinine to 2 times or more from baseline within 7 to 90 days.
3. Post-discharge estimated glomerular filtration rate (eGFR) between 30 and 60 ml/min/1.73m², calculated using the MDRD equation.
4. Hospitalization duration not exceeding 1 month.

Exclusion criteria

1. Patients with cancer or hematological malignancies.
2. Patients with AKD etiologies that cannot be managed in an outpatient setting (e.g., diabetic foot, obstructive uropathy with sepsis, cirrhosis).

1. Patients presenting any of the following conditions, considered as excessively vulnerable populations or other conditions:

* Bedridden.
* Requiring nasogastric tube feeding.
* Long-term use of oxygen therapy.
* Use of urinary catheters.

Patients unsuitable for AST-120 treatment, including:

* Patients with severe constipation (defined as requiring the daily use of more than one laxative).
* Patients with abnormal liver function (defined as ALT levels greater than 5 times the upper limit or total bilirubin > 2mg/dL).
* Patients with a history of peptic ulcers within the last month.
* Pregnant women.
* Patients allergic to the study drug.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-02-11 (Estimated); Study Completion 2027-03-13 (Estimated)

PRIMARY OUTCOMES:
Change in serum indoxyl sulfate (IS) concentration | Day 0, Day 14, Day 90, Day 180
  Change in serum indoxyl sulfate (IS) concentration
  Time Frame: Baseline to Day 180
  Description: Evaluate reduction in IS levels after AST-120 treatment compared to control.

SECONDARY OUTCOMES:
Change in serum p-cresyl sulfate (p-CS) concentration | Day 0, Day 14, Day 90, Day 180
  Change in serum p-cresyl sulfate (p-CS) concentration Time Frame: Baseline to Day 180 Assess difference in p-CS levels between groups.
Change in estimated glomerular filtration rate (eGFR) | Day 0, Day 14, Day 90, Day 180
  Change in estimated glomerular filtration rate (eGFR) Time Frame: Baseline to Day 180 Description: Evaluate reduction in eGFR after AST-120 treatment compared to control.
Change in urine albumin/creatinine ratio (UACR) | Day 0, Day 14, Day 90, Day 180
  Change in urine albumin/creatinine ratio (UACR)
  Time Frame: Baseline to Day 180
  Description: Evaluate reduction inUACR after AST-120 treatment compared to control.
Change in urine total protein/creatinine ratio (UPCR) | Day 0, Day 14, Day 90, Day 180
  Change in urine total protein/creatinine ratio (UPCR) Time Frame: Baseline to Day 180 Description: Evaluate reduction in UPCR after AST-120 treatment compared to control.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan, Taiwan, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caillard P, Bennis Y, Six I, Bodeau S, Kamel S, Choukroun G, Maizel J, Titeca-Beauport D. The Role of Gut-Derived, Protein-Bound Uremic Toxins in the Cardiovascular Complications of Acute Kidney Injury. Toxins (Basel). 2022 May 11;14(5):336. doi: 10.3390/toxins14050336. PMID 35622583
- [Background] Yamamoto S, Kazama JJ, Omori K, Matsuo K, Takahashi Y, Kawamura K, Matsuto T, Watanabe H, Maruyama T, Narita I. Continuous Reduction of Protein-Bound Uraemic Toxins with Improved Oxidative Stress by Using the Oral Charcoal Adsorbent AST-120 in Haemodialysis Patients. Sci Rep. 2015 Sep 23;5:14381. doi: 10.1038/srep14381. PMID 26395517
- [Background] Nagata D, Yoshizawa H. Pharmacological Actions of Indoxyl Sulfate and AST-120 That Should Be Recognized for the Strategic Treatment of Patients with Chronic Kidney Disease. Int J Nephrol Renovasc Dis. 2020 Dec 4;13:359-365. doi: 10.2147/IJNRD.S287237. eCollection 2020. PMID 33311993
- [Background] Shen WC, Chou YH, Shi LS, Chen ZW, Tu HJ, Lin XY, Wang GJ. AST-120 Improves Cardiac Dysfunction in Acute Kidney Injury Mice via Suppression of Apoptosis and Proinflammatory NF-kappaB/ICAM-1 Signaling. J Inflamm Res. 2021 Feb 24;14:505-518. doi: 10.2147/JIR.S283378. eCollection 2021. PMID 33658826
- [Background] Lim YJ, Sidor NA, Tonial NC, Che A, Urquhart BL. Uremic Toxins in the Progression of Chronic Kidney Disease and Cardiovascular Disease: Mechanisms and Therapeutic Targets. Toxins (Basel). 2021 Feb 13;13(2):142. doi: 10.3390/toxins13020142. PMID 33668632
- [Background] Espi M, Koppe L, Fouque D, Thaunat O. Chronic Kidney Disease-Associated Immune Dysfunctions: Impact of Protein-Bound Uremic Retention Solutes on Immune Cells. Toxins (Basel). 2020 May 6;12(5):300. doi: 10.3390/toxins12050300. PMID 32384617
- [Background] Schulman G, Berl T, Beck GJ, Remuzzi G, Ritz E, Arita K, Kato A, Shimizu M. Randomized Placebo-Controlled EPPIC Trials of AST-120 in CKD. J Am Soc Nephrol. 2015 Jul;26(7):1732-46. doi: 10.1681/ASN.2014010042. Epub 2014 Oct 27. PMID 25349205
- [Background] Sun CY, Chang SC, Wu MS. Suppression of Klotho expression by protein-bound uremic toxins is associated with increased DNA methyltransferase expression and DNA hypermethylation. Kidney Int. 2012 Apr;81(7):640-50. doi: 10.1038/ki.2011.445. Epub 2012 Jan 11. PMID 22237753
- [Background] Chen JH, Chiang CK. Uremic Toxins and Protein-Bound Therapeutics in AKI and CKD: Up-to-Date Evidence. Toxins (Basel). 2021 Dec 23;14(1):8. doi: 10.3390/toxins14010008. PMID 35050985
- [Background] Sun CY, Hsu HH, Wu MS. p-Cresol sulfate and indoxyl sulfate induce similar cellular inflammatory gene expressions in cultured proximal renal tubular cells. Nephrol Dial Transplant. 2013 Jan;28(1):70-8. doi: 10.1093/ndt/gfs133. Epub 2012 May 18. PMID 22610984
- [Background] Barreto FC, Barreto DV, Liabeuf S, Meert N, Glorieux G, Temmar M, Choukroun G, Vanholder R, Massy ZA; European Uremic Toxin Work Group (EUTox). Serum indoxyl sulfate is associated with vascular disease and mortality in chronic kidney disease patients. Clin J Am Soc Nephrol. 2009 Oct;4(10):1551-8. doi: 10.2215/CJN.03980609. Epub 2009 Aug 20. PMID 19696217
- [Background] Schulman G, Vanholder R, Niwa T. AST-120 for the management of progression of chronic kidney disease. Int J Nephrol Renovasc Dis. 2014 Jan 30;7:49-56. doi: 10.2147/IJNRD.S41339. eCollection 2014. PMID 24501542
- [Background] Levey AS. Defining AKD: The Spectrum of AKI, AKD, and CKD. Nephron. 2022;146(3):302-305. doi: 10.1159/000516647. Epub 2021 Jun 24. PMID 34167119